CLINICAL TRIAL: NCT02763527
Title: The Effectiveness of Negotiating Self-Determination to Reduce Cigarette Consumption (NSD-RCC) Among Smokers Attending Outpatient Clinics: A Cluster Randomized Controlled Trial
Brief Title: Effectiveness of Negotiating Self-determination to Reduce Cigarette Consumption
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GRF
Record Dates: First submitted 2016-04-26; First posted 2016-05-05 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Smoking
Keywords: smoking cessation
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoking reduction (Experimental): Subjects will receive a brief intervention on smoking reduction with a warning message plus a smoking reduction leaflet. They will be asked to think about a tailored smoking reduction schedule for themselves after the negotiation with the trained counsellor. The trained counsellor will negotiate a schedule with subjects to reduce their smoking over an acceptable level. For the subsequent telephone follow up in the intervention group, information on reduction and cessation will be collected, followed by a "booster" intervention, which will repeat the health warning to positively encourage them to reinforce their efforts and the next reduction target. Four consecutive (1, 3, 6 and 12 months) follow-ups will be conducted over the telephone by trained interviewers.
  Interventions: Behavioral: Smoking reduction
- Smoking Cessation (Placebo Comparator): Subjects in the QI group will always be advised to quit immediately rather than to quit progressively. Subjects will receive a brief advice on quitting with a warning message similar to subjects in the QP group. In addition, subjects will receive a self-help quitting pamphlet published by the Hong Kong Council on Smoking and Health (COSH). Unlike the QP group, subjects in the QI group will not receive smoking reduction intervention and leaflet, and "booster" intervention during telephone follow-ups. However, they will undergo a similar schedule of telephone follow-up as those in the QP group.
  Interventions: Behavioral: Smoking Cessation

INTERVENTIONS:
Behavioral: Smoking reduction — A brief intervention on smoking reduction plus a smoking reduction leaflet
  Arms: Smoking reduction
Behavioral: Smoking Cessation — A brief advice on quitting plus a leaflet on smoking cessation
  Arms: Smoking Cessation

SUMMARY:
Background: Smokers attended to outpatient clinics present an excellent 'teachable moment' for smoking cessation interventions. This protocol paper describes the rationale and methods of a large randomized controlled trial which aims to evaluate the effectiveness of negotiating self-determination to reduce cigarette consumption among smokers attending outpatient clinics

Methods: A randomized controlled trial will be conducted in 10 out-patient clinics in Hong Kong. Subjects in the intervention group will receive a brief intervention on smoking reduction plus a smoking reduction leaflet. Additionally, subjects will be asked to think about a smoking reduction schedule for themselves after the negotiation with the counsellor. Subjects in the control group will receive a brief advice on quitting plus a leaflet on smoking cessation. Four consecutive (1, 3, 6 and 12 months) follow-ups will be conducted. The primary outcome measure is biochemically validated abstinence at 6 months. Secondary outcomes are: (i) biochemically validated abstinence at 12 months, (ii) self-reported 7-day point prevalence of abstinence at 6 and 12 months, (iii) self-reported reduction of ≥ 50% in cigarette consumption at 6 and 12 months, and (iv) self-efficacy against tobacco at 6 and 12 months.

DETAILED DESCRIPTION:
This study aims to test the effectiveness of negotiating self-determination to reduce cigarette consumption (NSD-RCC) among smokers attending outpatient clinics.

Intervention Group (QP) Subjects in this group will receive a brief intervention on smoking reduction with a warning message plus a smoking reduction leaflet (the content will include a roadmap of smoking reduction strategy and information on how to cope with nicotine withdrawal symptoms). The whole intervention will last about 1 minute or slightly longer if necessary. In addition, subjects will be asked to think about a tailored smoking reduction schedule for themselves after the negotiation with the trained counsellor. For the subsequent telephone follow up in the intervention group, information on reduction and cessation will be collected, followed by a "booster" intervention, which will repeat the health warning to positively encourage them to reinforce their efforts and the next reduction target.

Control Group (QI) Subjects in the QI group will always be advised to quit immediately rather than to quit progressively. Subjects will receive a brief advice on quitting with a warning message similar to subjects in the QP group. In addition, subjects will receive a self-help quitting pamphlet published by the Hong Kong Council on Smoking and Health (COSH). Unlike the QP group, subjects in the QI group will not receive smoking reduction intervention and leaflet, and "booster" intervention during telephone follow-ups. However, they will undergo a similar schedule of telephone follow-up as those in the QP group.

Data collection

After completing the baseline questionnaire, subjects will receive proposed intervention according to their group assignment. Four consecutive follow-ups (at 1, 3, 6 and 12 months) will be conducted over the telephone by trained interviewers. Interviewers will first carry out outcome assessments with blinding to group status. Then, the group status will be disclosed so that the intervention group will receive the booster intervention and the control group will not. Smokers who have successfully quit smoking at 6-month will be invited to come back to the out-patient clinic and have biochemical validation tests (saliva cotinine test and exhaled CO test).

Analysis Data analysis will be performed using the Statistical Package for Social Science. We will compare the baseline characteristics of the participants by chi-square test for categorical variables and F-test for continuous variables between the intervention and the control group. We shall use the chi-square test to assess the effect of intervention and calculate the crude odds ratio (OR) with 95% confidence interval (CI) for the primary and secondary outcomes. Those who are lost to follow-up or refuse to participate in the validation tests, will be treated as smokers with no reduction in cigarette consumption compared with (a) baseline, as the main analysis (by intention to treat), (b) the most recent level and (c) complete case (per protocol) analysis by excluding subjects with missing data as a sensitivity analysis.

ELIGIBILITY:
Inclusion Criteria:

smokers

* who are Chinese
* aged 18 years or above
* who smoke at least two cigarettes per day
* with moderate to severe nicotine dependence, and
* have no intention to quit smoking ≤7 days, but are interested in reducing the number of cigarettes smoked per day .

Exclusion Criteria:

smokers

* with unstable medical conditions as advised by the doctor in charge,
* with poor cognitive state or mental illness,
* who participate in other smoking cessation programmes or services,
* with mild nicotine dependence, or
* who claim that they can quit ≤7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1566 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
biochemically validated abstinence using exhaled CO test | 6 months

SECONDARY OUTCOMES:
biochemically validated abstinence using exhaled CO test | 12 months
self-reported 7-day point prevalence of abstinence | 6 months
self-reported 7-day point prevalence of abstinence | 12 months
self-reported reduction of ≥ 50% in cigarette consumption | 6 months
self-reported reduction of ≥ 50% in cigarette consumption | 12 months
self-efficacy against tobacco | 6 months
  Subjects' self-efficacy against tobacco was assessed by using 12-item Smoking Self-efficacy Questionnaire (SEQ-12). SEQ-12 is a valid and reliable scale, which has been used in both research and clinical setting.
self-efficacy against tobacco | 12 months
  Subjects' self-efficacy against tobacco was assessed by using 12-item Smoking Self-efficacy Questionnaire (SEQ-12). SEQ-12 is a valid and reliable scale, which has been used in both research and clinical setting.
biochemically validated abstinence using saliva cotinine test | 6 months
biochemically validated abstinence using saliva cotinine test | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: William, Ho Cheung LI, PhD, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No